CLINICAL TRIAL: NCT04356001
Title: The "One-piece" Autologous Tuberosity Graft : a Novel Concept in Ridge Preservation
Brief Title: The "One-piece" Autologous Tuberosity Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USJ -2018-65
Record Dates: First submitted 2020-03-06; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: extraction; socket preservation; autologous; maxillary tuberosity; hard and soft tissue graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Socket preservation group (Experimental): Extraction sockets filled with a "one-piece" dual tissue graft harvested from the tuberosity using an adjusted trephine.
  Interventions: Procedure: Socket preservation

INTERVENTIONS:
Procedure: Socket preservation — 'One-Piece' autologous tuberosity graft combining hard and soft tissue, harvested from the maxillary tuberosity, placed in extraction sockets.
  Other Names: autologous tuberosity graft

SUMMARY:
A prospective study investigating clinically and radiologically the effectiveness of the use of a combined hard and soft tissue graft retrieved from the maxillary tuberosity and designed for alveolar ridge preservation following tooth extraction.

DETAILED DESCRIPTION:
Patients scheduled for a single mono-rooted tooth extraction are included in the study. After atraumatic extraction, sockets are filled with a "one-piece" dual tissue graft harvested from the tuberosity using an adjusted trephine. CBCTs are performed before the extraction and 4 months after ridge preservation, to analyze the vertical and horizontal alterations of the ridge, using 'ITK-Snap' software.

Clinical measurements of both soft and hard tissues are also assessed during the extraction and implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient
* Patient with at least one single-rooted tooth to be extracted and be replaced with an implant
* No signs of acute infection : edema, suppuration, abscess, spontaneous bleeding
* Non-smoker or Light Smoker < 10 cigarettes/day

Exclusion Criteria:

* Pregnant or lactating females
* Non-controlled periodontal disease
* Medical conditions that contraindicate implant surgery
* Metabolic bone disorders such as osteoporosis,..
* Severe psychiatric conditions
* Heavy smoker > 10 cigarettes/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Change of volume of the ridge from baseline to 4 months post-op | 4 months
  Volumetric variation of the ridge, measured on superimposed images of CBCT.
Change of Vertical dimension of the ridge from baseline to 4 months post-op | 4 months
  Linear Vertical variation of the ridge, measured on superimposed images of CBCT.
Change of Horizontal dimension of the ridge from baseline to 4 months post-op | 4 months
  Linear Horizontal variation of the ridge at 3 different levels, measured on superimposed images of CBCT.
Change in Soft tissue from baseline to 4 months post-op | 4 months
  Variation of the thickness of the buccal keratinized mucosa at 2 different levels, measured on superimposed images of CBCT.

SECONDARY OUTCOMES:
Change in buccal Soft tissue from baseline to 4 months post-op (clinical measurements) | 4 months
  Thickness of the keratinized mucosa on the buccal site, measured with a gauge caliper.
Change in crestal Soft tissue from baseline to 4 months post-op (clinical measurements) | 4 months
  Thickness of the keratinized mucosa on the crestal site, measured with a gauge caliper.
Change in Hard tissue from baseline to 4 months post-op (clinical measurements) | 4 months
  Horizontal dimension of the ridge (bucco-lingual) measured with a periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Joseph university, Beirut, Lebanon